CLINICAL TRIAL: NCT00005275
Title: The Sleep Heart Health Study (SHHS) Was a Multi-site Prospective Cohort Study to Investigate Obstructive Sleep Apnea (OSA) and Other Sleep-disordered Breathing (SDB) as Risk Factors for Cardiovascular Diseases and Hypertension
Brief Title: Sleep Heart Health Study (SHHS) Data Coordinating Center
Acronym: SHHS
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marie Diener-West, Professor, Johns Hopkins Bloomberg School of Public Health
Other Study IDs: 1302; U01HL053941-14 (NIH); U01HL053941 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Lung Diseases; Sleep Apnea Syndromes; Cardiovascular Diseases; Heart Diseases; Coronary Disease; Cerebrovascular Accident; Hypertension; Myocardial Infarction
MeSH Terms: conditions — Lung Diseases; Sleep Apnea Syndromes; Cardiovascular Diseases; Heart Diseases; Coronary Disease; Stroke; Hypertension; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To test whether sleep-disordered breathing is associated with an increased risk of coronary heart disease, stroke, all-cause mortality, and hypertension. The multicenter, longitudinal study draws on existing, well-characterized, and established epidemiologic cohorts.

DETAILED DESCRIPTION:
BACKGROUND:

The study was motivated by the increasing recognition of the frequent occurrences of sleep-disordered breathing in the general population and mounting evidence that sleep-disordered breathing may increase risk for cardiovascular diseases, including coronary artery disease and stroke, and for hypertension, and may reduce quality of life generally. Many clinical questions remain unanswered concerning sleep-disordered breathing as well: for example, when, in the natural history of the disorder, intervention is warranted; and how to determine who is at risk so that recently developed treatments can be applied in a cost-effective manner.

The initiative was developed by the Pulmonary Diseases Advisory Committee, approved by the full Committee in February, 1993, and given concept clearance by the October, 1993 National Heart, Lung, and Blood Advisory Council. The Request for Applications was released in January, 1994.

DESIGN NARRATIVE:

The SHHS adds in-home polysomnography to the data collected in each of the cohorts under study. Using the Compumedics SleepWatch polysomnograph, a single over-night polysomnogram is obtained at home for the subjects; the montage includes oximetry, heart rate, chest wall and abdominal movement, nasal/oral airflow, body position, EEG, ECG, and chin EMG. In-home monitoring provides data on the occurrence of sleep-disordered breathing and on arousals.

Although the SHHS is a prospective cohort study, the cross-sectional findings will provide new information on patterns of sleep and sleep-disordered breathing in the general population. Consequently, initial analyses will be descriptive and will also address cross-sectional associations of sleep-disordered breathing with prevalent cardiovascular disease and quality of life and with risk factors for cardiovascular disease. Longitudinal analyses will address sleep-disordered breathing as a predictor of cardiovascular outcomes and change in blood pressure.

The extent of information available on key cardiovascular risk factors varies among the parent cohorts. Some additional data are collected on covariates at enrollment into the SHHS. However, the parent studies are the principal source of information on risk factors for cardiovascular disease in the participants. The cardiovascular outcomes for all sites include hospitalized acute myocardial infarction, nonfatal coronary heart disease, stroke, and death due to cardiovascular or cerebrovascular disease. Change in blood pressure and diagnosis of hypertension is considered, and all participants complete a standardized instrument on quality of life. The cardiovascular outcomes are adjudicated by methods already in place for the ARIC, CHS, SHS, and Framingham Field Centers and by the CHS process for the New York and Tucson Field Centers. Ancillary studies address other outcomes, such as cognitive functioning, that cannot be considered in the full SHHS cohort.

STATUS:

Over 80 manuscripts were published based on substudies and ancillary investigations. Three primary outcomes papers were published in 2009 and 2010, based on follow-up as of 2006-2007.

The study was renewed several times to provide for continued data collection and follow-up, including new polysomnograms. The formal funding for SHHS sites, which ended as of August 31, 2008, was followed by a one-year no- cost extension. Funding ceased for the participating sites as of August 31, 2009, but the Data Coordinating Center and the PSG Reading Center were granted additional no-cost extensions to support additional data collection from the parent cohorts to obtain follow up through 2009, 2010 or 2011 (depending on the cohort), on all-cause mortality, incident CVD, and stroke. The updated results were presented in a session at the ATS 2012 meetings in San Francisco.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years and older
* Able and willing to undergo a home polysomnogram

Exclusion Criteria:

* Age < 40 years
* Unwillingness, or social, physical or mental condition precluding a home polysomnogram

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in SHHS were recruited from NHLBI cohort studies already in progress. Parent cohort studies and recruitment targets for these cohorts were as follows:
  * Atherosclerosis Risk in Communities Study (ARIC) - 1,750 participants
  * Cardiovascular Health Study (CHS) - 1,350 participants
  * Framingham Heart Study (FHS) - 1,000 participants
  * Strong Heart Study (SHS) - 600 participants
  * New York Hypertension Cohorts - 1,000 participants
  * Tucson Epidemiologic Study of Airways Obstructive Diseases and the Health and Environment Study - 900 participants
Sampling Method: Non-Probability Sample
Enrollment: 6441 (Actual)
Dates: Start 1994-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | 1998-2011
  Mortality subsequent to polysomnography performed in phase 1(1998-2000) for 6441 participants and in phase 2 (2001-2003) for 4381 participants. The latest follow-up data were collected from the parent cohorts in 2009-2011.

OTHER OUTCOMES:
Prevalent cardiovascular events and stroke | 1998-2011

CONTACTS AND LOCATIONS:
Overall Officials: George O'Connor, MD, MS, Principal Investigator — Boston University; Naresh Punjabi, MD, PhD, Principal Investigator — Johns Hopkins University; Stuart Quan, MD, Study Chair — Harvard Medical School (HMS and HSDM); David Rapoport, MD, Principal Investigator — NYU Langone Health; Susan Redline, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Helaine Resnick, PhD, Principal Investigator — Leading Age; John Robbins, MD, Principal Investigator — University of California, Davis; Jonathan Samet, MD, MS, Principal Investigator — University of Southern California; Eyal Shahar, MD, MPH, Principal Investigator — University of Arizona; Marie Diener-West, PhD, Principal Investigator — Johns Hopkins University; Anne Newman, MD, MPH, Principal Investigator — University of Pittsburgh

REFERENCES:
- [Background] Redline S, Sanders MH, Lind BK, Quan SF, Iber C, Gottlieb DJ, Bonekat WH, Rapoport DM, Smith PL, Kiley JP. Methods for obtaining and analyzing unattended polysomnography data for a multicenter study. Sleep Heart Health Research Group. Sleep. 1998 Nov 1;21(7):759-67. PMID 11300121
- [Background] Whitney CW, Gottlieb DJ, Redline S, Norman RG, Dodge RR, Shahar E, Surovec S, Nieto FJ. Reliability of scoring respiratory disturbance indices and sleep staging. Sleep. 1998 Nov 1;21(7):749-57. doi: 10.1093/sleep/21.7.749. PMID 11286351
- [Background] Gottlieb DJ, Whitney CW, Bonekat WH, Iber C, James GD, Lebowitz M, Nieto FJ, Rosenberg CE. Relation of sleepiness to respiratory disturbance index: the Sleep Heart Health Study. Am J Respir Crit Care Med. 1999 Feb;159(2):502-7. doi: 10.1164/ajrccm.159.2.9804051. PMID 9927364
- [Background] Quan SF, Howard BV, Iber C, Kiley JP, Nieto FJ, O'Connor GT, Rapoport DM, Redline S, Robbins J, Samet JM, Wahl PW. The Sleep Heart Health Study: design, rationale, and methods. Sleep. 1997 Dec;20(12):1077-85. PMID 9493915
- [Background] Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, D'Agostino RB, Newman AB, Lebowitz MD, Pickering TG. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA. 2000 Apr 12;283(14):1829-36. doi: 10.1001/jama.283.14.1829. PMID 10770144
- [Background] Whitney CW, Lind BK, Wahl PW. Quality assurance and quality control in longitudinal studies. Epidemiol Rev. 1998;20(1):71-80. doi: 10.1093/oxfordjournals.epirev.a017973. PMID 9762510
- [Background] Redline S, Sanders M. Hypopnea, a floating metric: implications for prevalence, morbidity estimates, and case finding. Sleep. 1997 Dec;20(12):1209-17. doi: 10.1093/sleep/20.12.1209. PMID 9493935
- [Background] Redline S, Kapur VK, Sanders MH, Quan SF, Gottlieb DJ, Rapoport DM, Bonekat WH, Smith PL, Kiley JP, Iber C. Effects of varying approaches for identifying respiratory disturbances on sleep apnea assessment. Am J Respir Crit Care Med. 2000 Feb;161(2 Pt 1):369-74. doi: 10.1164/ajrccm.161.2.9904031. PMID 10673173
- [Background] Shahar E, Whitney CW, Redline S, Lee ET, Newman AB, Nieto FJ, O'Connor GT, Boland LL, Schwartz JE, Samet JM. Sleep-disordered breathing and cardiovascular disease: cross-sectional results of the Sleep Heart Health Study. Am J Respir Crit Care Med. 2001 Jan;163(1):19-25. doi: 10.1164/ajrccm.163.1.2001008. PMID 11208620
- [Background] Baldwin CM, Griffith KA, Nieto FJ, O'Connor GT, Walsleben JA, Redline S. The association of sleep-disordered breathing and sleep symptoms with quality of life in the Sleep Heart Health Study. Sleep. 2001 Feb 1;24(1):96-105. doi: 10.1093/sleep/24.1.96. PMID 11204058
- [Background] Newman AB, Nieto FJ, Guidry U, Lind BK, Redline S, Pickering TG, Quan SF; Sleep Heart Health Study Research Group. Relation of sleep-disordered breathing to cardiovascular disease risk factors: the Sleep Heart Health Study. Am J Epidemiol. 2001 Jul 1;154(1):50-9. doi: 10.1093/aje/154.1.50. PMID 11434366
- [Background] Kapur VK, Rapoport DM, Sanders MH, Enright P, Hill J, Iber C, Romaniuk J. Rates of sensor loss in unattended home polysomnography: the influence of age, gender, obesity, and sleep-disordered breathing. Sleep. 2000 Aug 1;23(5):682-8. PMID 10947036
- [Background] Gottlieb DJ, Yao Q, Redline S, Ali T, Mahowald MW. Does snoring predict sleepiness independently of apnea and hypopnea frequency? Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1512-7. doi: 10.1164/ajrccm.162.4.9911073. PMID 11029370
- [Background] Young T, Shahar E, Nieto FJ, Redline S, Newman AB, Gottlieb DJ, Walsleben JA, Finn L, Enright P, Samet JM; Sleep Heart Health Study Research Group. Predictors of sleep-disordered breathing in community-dwelling adults: the Sleep Heart Health Study. Arch Intern Med. 2002 Apr 22;162(8):893-900. doi: 10.1001/archinte.162.8.893. PMID 11966340
- [Background] Kapur VK, Redline S, Nieto FJ, Young TB, Newman AB, Henderson JA; Sleep Heart Health Research Group. The relationship between chronically disrupted sleep and healthcare use. Sleep. 2002 May 1;25(3):289-96. PMID 12003159
- [Background] Boland LL, Shahar E, Iber C, Knopman DS, Kuo TF, Nieto FJ; Sleep Heart Health Study (SHHS) Investigators. Measures of cognitive function in persons with varying degrees of sleep-disordered breathing: the Sleep Heart Health Study. J Sleep Res. 2002 Sep;11(3):265-72. doi: 10.1046/j.1365-2869.2002.00308.x. PMID 12220323
- [Background] Sanders MH, Newman AB, Haggerty CL, Redline S, Lebowitz M, Samet J, O'Connor GT, Punjabi NM, Shahar E; Sleep Heart Health Study. Sleep and sleep-disordered breathing in adults with predominantly mild obstructive airway disease. Am J Respir Crit Care Med. 2003 Jan 1;167(1):7-14. doi: 10.1164/rccm.2203046. PMID 12502472
- [Background] Resnick HE, Redline S, Shahar E, Gilpin A, Newman A, Walter R, Ewy GA, Howard BV, Punjabi NM; Sleep Heart Health Study. Diabetes and sleep disturbances: findings from the Sleep Heart Health Study. Diabetes Care. 2003 Mar;26(3):702-9. doi: 10.2337/diacare.26.3.702. PMID 12610025
- [Background] Quan SF, Griswold ME, Iber C, Nieto FJ, Rapoport DM, Redline S, Sanders M, Young T; Sleep Heart Health Study (SHHS) Research Group. Short-term variability of respiration and sleep during unattended nonlaboratory polysomnography--the Sleep Heart Health Study. [corrected]. Sleep. 2002 Dec;25(8):843-9. PMID 12489889
- [Background] Shahar E, Redline S, Young T, Boland LL, Baldwin CM, Nieto FJ, O'Connor GT, Rapoport DM, Robbins JA. Hormone replacement therapy and sleep-disordered breathing. Am J Respir Crit Care Med. 2003 May 1;167(9):1186-92. doi: 10.1164/rccm.200210-1238OC. Epub 2003 Jan 16. PMID 12531779
- [Background] Lind BK, Goodwin JL, Hill JG, Ali T, Redline S, Quan SF. Recruitment of healthy adults into a study of overnight sleep monitoring in the home: experience of the Sleep Heart Health Study. Sleep Breath. 2003 Mar;7(1):13-24. doi: 10.1007/s11325-003-0013-z. PMID 12712393
- [Background] O'Connor GT, Lind BK, Lee ET, Nieto FJ, Redline S, Samet JM, Boland LL, Walsleben JA, Foster GL; Sleep Heart Health Study Investigators. Variation in symptoms of sleep-disordered breathing with race and ethnicity: the Sleep Heart Health Study. Sleep. 2003 Feb 1;26(1):74-9. PMID 12627736
- [Background] Nieto FJ, Herrington DM, Redline S, Benjamin EJ, Robbins JA. Sleep apnea and markers of vascular endothelial function in a large community sample of older adults. Am J Respir Crit Care Med. 2004 Feb 1;169(3):354-60. doi: 10.1164/rccm.200306-756OC. Epub 2003 Oct 9. PMID 14551166
- [Background] Walsleben JA, Kapur VK, Newman AB, Shahar E, Bootzin RR, Rosenberg CE, O'Connor G, Nieto FJ. Sleep and reported daytime sleepiness in normal subjects: the Sleep Heart Health Study. Sleep. 2004 Mar 15;27(2):293-8. doi: 10.1093/sleep/27.2.293. PMID 15124725
- [Background] Kapur V, Strohl KP, Redline S, Iber C, O'Connor G, Nieto J. Underdiagnosis of sleep apnea syndrome in U.S. communities. Sleep Breath. 2002 Jun;6(2):49-54. doi: 10.1007/s11325-002-0049-5. PMID 12075479
- [Background] Iber C, Redline S, Kaplan Gilpin AM, Quan SF, Zhang L, Gottlieb DJ, Rapoport D, Resnick HE, Sanders M, Smith P. Polysomnography performed in the unattended home versus the attended laboratory setting--Sleep Heart Health Study methodology. Sleep. 2004 May 1;27(3):536-40. doi: 10.1093/sleep/27.3.536. PMID 15164911
- [Background] Boland LL, Shahar E, Wong TY, Klein R, Punjabi N, Robbins JA, Newman AB. Sleep-disordered breathing is not associated with the presence of retinal microvascular abnormalities: the Sleep Heart Health Study. Sleep. 2004 May 1;27(3):467-73. doi: 10.1093/sleep/27.3.467. PMID 15164900
- [Background] Redline S, Kirchner HL, Quan SF, Gottlieb DJ, Kapur V, Newman A. The effects of age, sex, ethnicity, and sleep-disordered breathing on sleep architecture. Arch Intern Med. 2004 Feb 23;164(4):406-18. doi: 10.1001/archinte.164.4.406. PMID 14980992
- [Background] Punjabi NM, Shahar E, Redline S, Gottlieb DJ, Givelber R, Resnick HE; Sleep Heart Health Study Investigators. Sleep-disordered breathing, glucose intolerance, and insulin resistance: the Sleep Heart Health Study. Am J Epidemiol. 2004 Sep 15;160(6):521-30. doi: 10.1093/aje/kwh261. PMID 15353412
- [Background] Gottlieb DJ, DeStefano AL, Foley DJ, Mignot E, Redline S, Givelber RJ, Young T. APOE epsilon4 is associated with obstructive sleep apnea/hypopnea: the Sleep Heart Health Study. Neurology. 2004 Aug 24;63(4):664-8. doi: 10.1212/01.wnl.0000134671.99649.32. PMID 15326239
- [Background] Valyi-Nagy I, Jensen PJ, Albelda SM, Rodeck U. Cytokine-induced expression of transforming growth factor-alpha and the epidermal growth factor receptor in neonatal skin explants. J Invest Dermatol. 1992 Sep;99(3):350-6. doi: 10.1111/1523-1747.ep12616672. PMID 1512472
- [Background] Haas DC, Foster GL, Nieto FJ, Redline S, Resnick HE, Robbins JA, Young T, Pickering TG. Age-dependent associations between sleep-disordered breathing and hypertension: importance of discriminating between systolic/diastolic hypertension and isolated systolic hypertension in the Sleep Heart Health Study. Circulation. 2005 Feb 8;111(5):614-21. doi: 10.1161/01.CIR.0000154540.62381.CF. PMID 15699282
- [Background] Ding J, Nieto FJ, Beauchamp NJ Jr, Harris TB, Robbins JA, Hetmanski JB, Fried LP, Redline S. Sleep-disordered breathing and white matter disease in the brainstem in older adults. Sleep. 2004 May 1;27(3):474-9. doi: 10.1093/sleep/27.3.474. PMID 15164901
- [Background] Gottlieb DJ, Punjabi NM, Newman AB, Resnick HE, Redline S, Baldwin CM, Nieto FJ. Association of sleep time with diabetes mellitus and impaired glucose tolerance. Arch Intern Med. 2005 Apr 25;165(8):863-7. doi: 10.1001/archinte.165.8.863. PMID 15851636
- [Background] Fass R, Quan SF, O'Connor GT, Ervin A, Iber C. Predictors of heartburn during sleep in a large prospective cohort study. Chest. 2005 May;127(5):1658-66. doi: 10.1378/chest.127.5.1658. PMID 15888843
- [Background] Levy AP, Zhang L, Miller-Lotan R, Redline S, O'Connor GT, Quan SF, Resnick HE. Haptoglobin phenotype, sleep-disordered breathing, and the prevalence of cardiovascular disease: the Sleep Heart Health Study. Sleep. 2005 Feb;28(2):207-13. doi: 10.1093/sleep/28.2.207. PMID 16171245
- [Background] Newman AB, Foster G, Givelber R, Nieto FJ, Redline S, Young T. Progression and regression of sleep-disordered breathing with changes in weight: the Sleep Heart Health Study. Arch Intern Med. 2005 Nov 14;165(20):2408-13. doi: 10.1001/archinte.165.20.2408. PMID 16287771
- [Background] Robbins J, Redline S, Ervin A, Walsleben JA, Ding J, Nieto FJ. Associations of sleep-disordered breathing and cerebral changes on MRI. J Clin Sleep Med. 2005 Apr 15;1(2):159-65. PMID 17561631
- [Background] Redline S, Min NI, Shahar E, Rapoport D, O'Connor G. Polysomnographic predictors of blood pressure and hypertension: is one index best? Sleep. 2005 Sep;28(9):1122-30. doi: 10.1093/sleep/28.9.1122. PMID 16268382
- [Background] Mehra R, Benjamin EJ, Shahar E, Gottlieb DJ, Nawabit R, Kirchner HL, Sahadevan J, Redline S; Sleep Heart Health Study. Association of nocturnal arrhythmias with sleep-disordered breathing: The Sleep Heart Health Study. Am J Respir Crit Care Med. 2006 Apr 15;173(8):910-6. doi: 10.1164/rccm.200509-1442OC. Epub 2006 Jan 19. PMID 16424443
- [Background] Gottlieb DJ, Redline S, Nieto FJ, Baldwin CM, Newman AB, Resnick HE, Punjabi NM. Association of usual sleep duration with hypertension: the Sleep Heart Health Study. Sleep. 2006 Aug;29(8):1009-14. doi: 10.1093/sleep/29.8.1009. PMID 16944668
- [Background] Quan SF, Wright R, Baldwin CM, Kaemingk KL, Goodwin JL, Kuo TF, Kaszniak A, Boland LL, Caccappolo E, Bootzin RR. Obstructive sleep apnea-hypopnea and neurocognitive functioning in the Sleep Heart Health Study. Sleep Med. 2006 Sep;7(6):498-507. doi: 10.1016/j.sleep.2006.02.005. Epub 2006 Jul 3. PMID 16815753
- [Background] Zhang L, Samet J, Caffo B, Punjabi NM. Cigarette smoking and nocturnal sleep architecture. Am J Epidemiol. 2006 Sep 15;164(6):529-37. doi: 10.1093/aje/kwj231. Epub 2006 Jul 7. PMID 16829553
- [Background] Patwardhan AA, Larson MG, Levy D, Benjamin EJ, Leip EP, Keyes MJ, Wang TJ, Gottlieb DJ, Vasan RS. Obstructive sleep apnea and plasma natriuretic peptide levels in a community-based sample. Sleep. 2006 Oct;29(10):1301-6. doi: 10.1093/sleep/29.10.1301. PMID 17068983
- [Background] Unruh ML, Sanders MH, Redline S, Piraino BM, Umans JG, Hammond TC, Sharief I, Punjabi NM, Newman AB. Sleep apnea in patients on conventional thrice-weekly hemodialysis: comparison with matched controls from the Sleep Heart Health Study. J Am Soc Nephrol. 2006 Dec;17(12):3503-9. doi: 10.1681/ASN.2006060659. Epub 2006 Nov 2. PMID 17082238
- [Background] Quan SF, O'Connor GT, Quan JS, Redline S, Resnick HE, Shahar E, Siscovick D, Sherrill DL. Association of physical activity with sleep-disordered breathing. Sleep Breath. 2007 Sep;11(3):149-57. doi: 10.1007/s11325-006-0095-5. PMID 17221274
- [Background] Wattanakit K, Boland L, Punjabi NM, Shahar E. Relation of sleep-disordered breathing to carotid plaque and intima-media thickness. Atherosclerosis. 2008 Mar;197(1):125-31. doi: 10.1016/j.atherosclerosis.2007.02.029. Epub 2007 Apr 11. PMID 17433330
- [Background] Gottlieb DJ, O'Connor GT, Wilk JB. Genome-wide association of sleep and circadian phenotypes. BMC Med Genet. 2007 Sep 19;8 Suppl 1(Suppl 1):S9. doi: 10.1186/1471-2350-8-S1-S9. PMID 17903308
- [Background] Zhang L, Samet J, Caffo B, Bankman I, Punjabi NM. Power spectral analysis of EEG activity during sleep in cigarette smokers. Chest. 2008 Feb;133(2):427-32. doi: 10.1378/chest.07-1190. Epub 2007 Oct 9. PMID 17925420
- [Background] Silva GE, Goodwin JL, Sherrill DL, Arnold JL, Bootzin RR, Smith T, Walsleben JA, Baldwin CM, Quan SF. Relationship between reported and measured sleep times: the sleep heart health study (SHHS). J Clin Sleep Med. 2007 Oct 15;3(6):622-30. PMID 17993045
- [Background] Winkelman JW, Shahar E, Sharief I, Gottlieb DJ. Association of restless legs syndrome and cardiovascular disease in the Sleep Heart Health Study. Neurology. 2008 Jan 1;70(1):35-42. doi: 10.1212/01.wnl.0000287072.93277.c9. PMID 18166705
- [Background] Seicean S, Kirchner HL, Gottlieb DJ, Punjabi NM, Resnick H, Sanders M, Budhiraja R, Singer M, Redline S. Sleep-disordered breathing and impaired glucose metabolism in normal-weight and overweight/obese individuals: the Sleep Heart Health Study. Diabetes Care. 2008 May;31(5):1001-6. doi: 10.2337/dc07-2003. Epub 2008 Feb 11. PMID 18268072
- [Background] Chami HA, Devereux RB, Gottdiener JS, Mehra R, Roman MJ, Benjamin EJ, Gottlieb DJ. Left ventricular morphology and systolic function in sleep-disordered breathing: the Sleep Heart Health Study. Circulation. 2008 May 20;117(20):2599-607. doi: 10.1161/CIRCULATIONAHA.107.717892. Epub 2008 May 5. PMID 18458174
- [Background] Punjabi NM, Newman AB, Young TB, Resnick HE, Sanders MH. Sleep-disordered breathing and cardiovascular disease: an outcome-based definition of hypopneas. Am J Respir Crit Care Med. 2008 May 15;177(10):1150-5. doi: 10.1164/rccm.200712-1884OC. Epub 2008 Feb 14. PMID 18276938
- [Background] Unruh ML, Redline S, An MW, Buysse DJ, Nieto FJ, Yeh JL, Newman AB. Subjective and objective sleep quality and aging in the sleep heart health study. J Am Geriatr Soc. 2008 Jul;56(7):1218-27. doi: 10.1111/j.1532-5415.2008.01755.x. Epub 2008 May 14. PMID 18482295
- [Background] Kapur VK, Resnick HE, Gottlieb DJ; Sleep Heart Health Study Group. Sleep disordered breathing and hypertension: does self-reported sleepiness modify the association? Sleep. 2008 Aug;31(8):1127-32. PMID 18714785
- [Background] Stamatakis K, Sanders MH, Caffo B, Resnick HE, Gottlieb DJ, Mehra R, Punjabi NM. Fasting glycemia in sleep disordered breathing: lowering the threshold on oxyhemoglobin desaturation. Sleep. 2008 Jul;31(7):1018-24. PMID 18652097
- [Background] Unruh ML, Sanders MH, Redline S, Piraino BM, Umans JG, Chami H, Budhiraja R, Punjabi NM, Buysse D, Newman AB. Subjective and objective sleep quality in patients on conventional thrice-weekly hemodialysis: comparison with matched controls from the sleep heart health study. Am J Kidney Dis. 2008 Aug;52(2):305-13. doi: 10.1053/j.ajkd.2008.04.019. Epub 2008 Jul 9. PMID 18617308
- [Background] Sharief I, Silva GE, Goodwin JL, Quan SF. Effect of sleep disordered breathing on the sleep of bed partners in the Sleep Heart Health Study. Sleep. 2008 Oct;31(10):1449-56. PMID 18853943
- [Background] O'Connor GT, Caffo B, Newman AB, Quan SF, Rapoport DM, Redline S, Resnick HE, Samet J, Shahar E. Prospective study of sleep-disordered breathing and hypertension: the Sleep Heart Health Study. Am J Respir Crit Care Med. 2009 Jun 15;179(12):1159-64. doi: 10.1164/rccm.200712-1809OC. Epub 2009 Mar 5. PMID 19264976
- [Background] Winkelman JW, Redline S, Baldwin CM, Resnick HE, Newman AB, Gottlieb DJ. Polysomnographic and health-related quality of life correlates of restless legs syndrome in the Sleep Heart Health Study. Sleep. 2009 Jun;32(6):772-8. doi: 10.1093/sleep/32.6.772. PMID 19544754
- [Background] Silva GE, An MW, Goodwin JL, Shahar E, Redline S, Resnick H, Baldwin CM, Quan SF. Longitudinal evaluation of sleep-disordered breathing and sleep symptoms with change in quality of life: the Sleep Heart Health Study (SHHS). Sleep. 2009 Aug;32(8):1049-57. doi: 10.1093/sleep/32.8.1049. PMID 19725256
- [Background] Chami HA, Keyes MJ, Vita JA, Mitchell GF, Larson MG, Fan S, Vasan RS, O'Connor GT, Benjamin EJ, Gottlieb DJ. Brachial artery diameter, blood flow and flow-mediated dilation in sleep-disordered breathing. Vasc Med. 2009 Nov;14(4):351-60. doi: 10.1177/1358863X09105132. PMID 19808720
- [Background] Monahan K, Storfer-Isser A, Mehra R, Shahar E, Mittleman M, Rottman J, Punjabi N, Sanders M, Quan SF, Resnick H, Redline S. Triggering of nocturnal arrhythmias by sleep-disordered breathing events. J Am Coll Cardiol. 2009 Nov 3;54(19):1797-804. doi: 10.1016/j.jacc.2009.06.038. PMID 19874994
- [Background] Caffo B, Swihart B, Laffan A, Crainiceanu C, Punjabi N. An overview of observational sleep research with application to sleep stage transitioning. Chance (N Y). 2009 Mar 1;22(1):10-15. doi: 10.1007/s144-009-0002-5. No abstract available. PMID 20046532
- [Background] Thomas RJ, Weiss MD, Mietus JE, Peng CK, Goldberger AL, Gottlieb DJ. Prevalent hypertension and stroke in the Sleep Heart Health Study: association with an ECG-derived spectrographic marker of cardiopulmonary coupling. Sleep. 2009 Jul;32(7):897-904. PMID 19639752
- [Background] Chami HA, Baldwin CM, Silverman A, Zhang Y, Rapoport D, Punjabi NM, Gottlieb DJ. Sleepiness, quality of life, and sleep maintenance in REM versus non-REM sleep-disordered breathing. Am J Respir Crit Care Med. 2010 May 1;181(9):997-1002. doi: 10.1164/rccm.200908-1304OC. Epub 2010 Jan 21. PMID 20093641
- [Background] Baldwin CM, Ervin AM, Mays MZ, Robbins J, Shafazand S, Walsleben J, Weaver T. Sleep disturbances, quality of life, and ethnicity: the Sleep Heart Health Study. J Clin Sleep Med. 2010 Apr 15;6(2):176-83. PMID 20411696
- [Background] Zanobetti A, Redline S, Schwartz J, Rosen D, Patel S, O'Connor GT, Lebowitz M, Coull BA, Gold DR. Associations of PM10 with sleep and sleep-disordered breathing in adults from seven U.S. urban areas. Am J Respir Crit Care Med. 2010 Sep 15;182(6):819-25. doi: 10.1164/rccm.200912-1797OC. Epub 2010 May 27. PMID 20508218
- [Background] Caffo B, Diener-West M, Punjabi NM, Samet J. A novel approach to prediction of mild obstructive sleep disordered breathing in a population-based sample: the Sleep Heart Health Study. Sleep. 2010 Dec;33(12):1641-8. doi: 10.1093/sleep/33.12.1641. PMID 21120126
- [Background] Larkin EK, Patel SR, Zhu X, Tracy RP, Jenny NS, Reiner AP, Walston J, Redline S. Study of the relationship between the interleukin-6 gene and obstructive sleep apnea. Clin Transl Sci. 2010 Dec;3(6):337-9. doi: 10.1111/j.1752-8062.2010.00236.x. PMID 21207764
- [Background] Laffan A, Caffo B, Swihart BJ, Punjabi NM. Utility of sleep stage transitions in assessing sleep continuity. Sleep. 2010 Dec;33(12):1681-6. doi: 10.1093/sleep/33.12.1681. PMID 21120130
- [Background] Chami HA, Resnick HE, Quan SF, Gottlieb DJ. Association of incident cardiovascular disease with progression of sleep-disordered breathing. Circulation. 2011 Mar 29;123(12):1280-6. doi: 10.1161/CIRCULATIONAHA.110.974022. Epub 2011 Mar 14. PMID 21403097
- [Background] Bruce EN, Bruce MC, Ramanand P, Hayes D Jr. Progressive changes in cortical state before and after spontaneous arousals from sleep in elderly and middle-aged women. Neuroscience. 2011 Feb 23;175:184-97. doi: 10.1016/j.neuroscience.2010.11.036. Epub 2010 Nov 27. PMID 21118712
- [Background] Silva GE, Vana KD, Goodwin JL, Sherrill DL, Quan SF. Identification of patients with sleep disordered breathing: comparing the four-variable screening tool, STOP, STOP-Bang, and Epworth Sleepiness Scales. J Clin Sleep Med. 2011 Oct 15;7(5):467-72. doi: 10.5664/JCSM.1308. PMID 22003341
- [Background] Parthasarathy S, Fitzgerald M, Goodwin JL, Unruh M, Guerra S, Quan SF. Nocturia, sleep-disordered breathing, and cardiovascular morbidity in a community-based cohort. PLoS One. 2012;7(2):e30969. doi: 10.1371/journal.pone.0030969. Epub 2012 Feb 6. PMID 22328924
- [Background] Budhiraja P, Budhiraja R, Goodwin JL, Allen RP, Newman AB, Koo BB, Quan SF. Incidence of restless legs syndrome and its correlates. J Clin Sleep Med. 2012 Apr 15;8(2):119-24. doi: 10.5664/jcsm.1756. PMID 22505854
- [Background] Aurora RN, Crainiceanu C, Caffo B, Punjabi NM. Sleep-disordered breathing and caffeine consumption: results of a community-based study. Chest. 2012 Sep;142(3):631-638. doi: 10.1378/chest.11-2894. PMID 22459776
- [Result] Punjabi NM, Caffo BS, Goodwin JL, Gottlieb DJ, Newman AB, O'Connor GT, Rapoport DM, Redline S, Resnick HE, Robbins JA, Shahar E, Unruh ML, Samet JM. Sleep-disordered breathing and mortality: a prospective cohort study. PLoS Med. 2009 Aug;6(8):e1000132. doi: 10.1371/journal.pmed.1000132. Epub 2009 Aug 18. PMID 19688045
- [Result] Redline S, Yenokyan G, Gottlieb DJ, Shahar E, O'Connor GT, Resnick HE, Diener-West M, Sanders MH, Wolf PA, Geraghty EM, Ali T, Lebowitz M, Punjabi NM. Obstructive sleep apnea-hypopnea and incident stroke: the sleep heart health study. Am J Respir Crit Care Med. 2010 Jul 15;182(2):269-77. doi: 10.1164/rccm.200911-1746OC. Epub 2010 Mar 25. PMID 20339144
- [Result] Gottlieb DJ, Yenokyan G, Newman AB, O'Connor GT, Punjabi NM, Quan SF, Redline S, Resnick HE, Tong EK, Diener-West M, Shahar E. Prospective study of obstructive sleep apnea and incident coronary heart disease and heart failure: the sleep heart health study. Circulation. 2010 Jul 27;122(4):352-60. doi: 10.1161/CIRCULATIONAHA.109.901801. Epub 2010 Jul 12. PMID 20625114
- [Derived] Martin-Montero A, Vaquerizo-Villar F, Garcia-Vicente C, Gutierrez-Tobal GC, Penzel T, Hornero R. Heart rate variability analysis in comorbid insomnia and sleep apnea (COMISA). Sci Rep. 2025 May 21;15(1):17574. doi: 10.1038/s41598-025-02541-7. PMID 40399494
- [Derived] Chen C, Guo Q, Cheng Y, Lan Y, Cheng D, Huang J. Naps and cardiovascular disease risk in different age and sex groups: evidence from a large community cohort. J Clin Sleep Med. 2024 Aug 1;20(8):1339-1348. doi: 10.5664/jcsm.11154. PMID 38607238
- [Derived] Morris JL, Scott PW, Magalang U, Keenan BT, Patel SR, Pack AI, Mazzotti DR. Five-year Transitions of Symptom Subtypes in Untreated Obstructive Sleep Apnea. medRxiv [Preprint]. 2023 May 19:2023.05.18.23290191. doi: 10.1101/2023.05.18.23290191. PMID 37292667
- [Derived] Zhao B, Meng Y, Jin X, Xi W, Ma Q, Yang J, Ma X, Yan B. Association of Objective and Self-Reported Sleep Duration With All-Cause and Cardiovascular Disease Mortality: A Community-Based Study. J Am Heart Assoc. 2023 Mar 21;12(6):e027832. doi: 10.1161/JAHA.122.027832. Epub 2023 Mar 9. PMID 36892074
- [Derived] Zhao B, Jin X, Yang J, Ma Q, Yang Z, Wang W, Bai L, Ma X, Yan B. Increased Rapid Eye Movement Sleep Is Associated With a Reduced Risk of Heart Failure in Middle-Aged and Older Adults. Front Cardiovasc Med. 2022 Mar 29;9:771280. doi: 10.3389/fcvm.2022.771280. eCollection 2022. PMID 35425819
- [Derived] Cho SE, Kang JM, Ko KP, Lim WJ, Redline S, Winkelman JW, Kang SG. Association Between Subjective-Objective Discrepancy of Sleeping Time and Health-Related Quality of Life: A Community-Based Polysomnographic Study. Psychosom Med. 2022 May 1;84(4):505-512. doi: 10.1097/PSY.0000000000001070. Epub 2022 Mar 23. PMID 35321997
- [Derived] Yan B, Wu Y, Fan X, Lu Q, Ma X, Bai L. Sleep fragmentation and incidence of congestive heart failure: the Sleep Heart Health Study. J Clin Sleep Med. 2021 Aug 1;17(8):1619-1625. doi: 10.5664/jcsm.9270. PMID 33779541
- [Derived] Yan B, Li J, Li R, Gao Y, Zhang J, Wang G. Association of daytime napping with incident cardiovascular disease in a community-based population. Sleep Med. 2019 May;57:128-134. doi: 10.1016/j.sleep.2019.02.014. Epub 2019 Mar 2. PMID 30981956
- [Derived] Zhang J, Jin X, Li R, Gao Y, Li J, Wang G. Influence of rapid eye movement sleep on all-cause mortality: a community-based cohort study. Aging (Albany NY). 2019 Mar 13;11(5):1580-1588. doi: 10.18632/aging.101858. PMID 30867337
- [Derived] Zhang J, Guo Q, Peng L, Li J, Gao Y, Yan B, Fang B, Wang G. The association of neck circumference with incident congestive heart failure and coronary heart disease mortality in a community-based population with or without sleep-disordered breathing. BMC Cardiovasc Disord. 2018 May 31;18(1):108. doi: 10.1186/s12872-018-0846-9. PMID 29855261